CLINICAL TRIAL: NCT00110240
Title: Efficacy and Safety of Vildagliptin Compared to Acarbose in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2323
Record Dates: First submitted 2005-05-04; First posted 2005-05-05 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This study is not being conducted in the United States. The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to acarbose in lowering overall blood glucose levels in people with type 2 diabetes who have not been previously treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Not currently on drug therapy for type 2 diabetes
* Body mass index (BMI) in the range 20-40
* Blood glucose criteria must be met

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of significant diabetic complications
* Evidence of serious cardiovascular conditions
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks

SECONDARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks for subset of Chinese patients
Overall adverse event profile after 24 weeks of treatment
Gastrointestinal side effect profiles after 24 weeks of treatment
Change from baseline in fasting plasma glucose at 24 weeks
Patients with endpoint HbA1c <7% after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Pan C, Yang W, Barona JP, Wang Y, Niggli M, Mohideen P, Wang Y, Foley JE. Comparison of vildagliptin and acarbose monotherapy in patients with Type 2 diabetes: a 24-week, double-blind, randomized trial. Diabet Med. 2008 Apr;25(4):435-41. doi: 10.1111/j.1464-5491.2008.02391.x. Epub 2008 Mar 13. PMID 18341596